CLINICAL TRIAL: NCT07053748
Title: Observational Clinical Study on High - Risk NMIBC Patients Choosing Trimodality Bladder - Sparing Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Shangbin QIN, Doctor, Peking University First Hospital
Other Study IDs: 2025-1081
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: High - Risk NMIBC
Keywords: Non-Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMT: High-risk NMIBC patients who have a strong desire to preserve their bladder actively choose to receive TMT bladder-preserving treatment instead of radical resection.
  Interventions: Radiation: Trimodality Bladder-preserving Therapy

INTERVENTIONS:
Radiation: Trimodality Bladder-preserving Therapy — High-risk NMIBC patients who have a strong desire to preserve their bladder actively choose to receive Trimodality Bladder-preserving Therapy instead of radical resection.

SUMMARY:
The goal of this observational study is to assess the safety and efficacy of trimodality bladder - sparing therapy in high - risk NMIBC patients. The main questions it aims to answer are:

Is trimodality therapy safe and effective in the short term for high - risk NMIBC patients? What is its long - term effectiveness in terms of EFS, OS, and BI - EFS? How does it affect patients' QOL? Participants will be high - risk NMIBC patients receiving trimodality therapy at Peking University First Hospital. They will be observed to evaluate the therapy's effectiveness and impact on QOL using relevant assessment criteria and QOL scores.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed NMIBC (Ta Tis T1).

≥2 recurrences after transurethral resection, or lack of response/intolerance to intravesical therapy (e.g., BCG).

Refusal of radical cystectomy and choice of TMT for bladder preservation. Aged ≥18 years. Signed informed consent. ECOG performance status of 0-2.

Adequate organ function for chemoradiotherapy:

Hematology: Absolute neutrophil count ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥90 g/L.

Liver function: Total bilirubin ≤1.5×ULN, ALT and AST ≤2.5×ULN (≤5×ULN if hepatic metastasis is present).

Renal function: Creatinine clearance ≥30 mL/min (via Cockcroft-Gault formula).

Exclusion Criteria:

Distant metastasis (M1). Other malignancies (except cured basal cell carcinoma or cervical carcinoma in situ).

Severe cardiovascular disease (uncontrolled heart failure, unstable angina, myocardial infarction, etc.).

Severe hepatic/renal dysfunction intolerance to chemoradiotherapy. Mental illness/cognitive impairment unable to comply with the study. Allergy to chemoradiotherapy drugs. Pregnant or breastfeeding women. Previous pelvic radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk patients with NMIBC who have a strong desire to preserve their bladder actively choose to receive TMT bladder treatment instead of radical resection.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
DFS | 5 years
OS | 5 Years
BI-DFS | 5 years